CLINICAL TRIAL: NCT00702481
Title: Phase II Study of Nimotuzumab (TheraCim-hR3) Concurrent With Cisplatin/Radiotherapy in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Study of Nimotuzumab and Cisplatin/Radiotherapy for Locally Advanced Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Innogene Kalbiotech Pte. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB/NCCS-01
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Squamous Cell Cancer; Chemoradiation; EGFR monoclonal antibody
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — nimotuzumab; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab/CDDP/RT (Experimental): Open label treatment arm of Nimotuzumab and cisplatin and radiation
  Interventions: Drug: Nimotuzumab; Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Nimotuzumab — Patients will receive nimotuzumab 200 mg weekly for 8 weeks. Nimotuzumab will be started together with concurrent chemoradiation, and continued 1 week after the completion of chemoradiation.
  Other Names: TheraCim-Rh3
Drug: Cisplatin — Concurrent chemotherapy with cisplatin 100 mg/m2 will be given on week 1, 4, and 7 of radiotherapy.
Radiation: Radiation — Concurrent radiotherapy will be given to the primary tumor and upper neck at 2 Gy per fraction, once a day, five days a week to a total of 70 Gy in 35 fractions in seven weeks.

SUMMARY:
The purpose of this study is to define the response and toxicities with the addition of Nimotuzumab to chemoradiation for head and neck cancer.

DETAILED DESCRIPTION:
Epidermal Growth Factor Receptor (EGFR) is overexpressed in Head and Neck Squamous Cell Carcinoma (HNSCC). EGFR pathway activation is associated with tumor growth, decreased apoptosis, and increased angiogenesis. These present a putative target for the use of EGFR inhibitors either in the form of small molecule inhibitors or monoclonal antibodies. Several studies have been advanced that suggest application of these targeted therapies show promising responses with little additional toxicity. The addition of EGFR monoclonal antibodies to radiation results in better response rates and locoregional control compared to radiation alone. Addition of EGFR monoclonal antibodies compared to chemotherapy alone also improves the response rates in patients with advanced HNSCC.

Nimotuzumab is a humanized chimeric monoclonal antibody specific to the extracellular domain of EGFR. Several studies are ongoing and demonstrate promising efficacy of Nimotuzumab as monotherapy and in combination with radiation in HNSCC, and in combination with chemoradiation in Nasopharyngeal Carcinoma. This phase II clinical trial examines the feasibility of EGFR inhibition using Nimotuzumab in combination with concurrent chemoradiotherapy in locally advanced unresectable HNSCC. Successful and safe incorporation of an EGFR monoclonal antibody into the concurrent chemoradiation paradigm used to treat locally advanced HNSCC will represent an important advance in the optimisation of treatment for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Squamous Cell Carcinoma of the Head and Neck.
* Locally advanced disease, unresectable disease or resectable disease where organ-preservation is intended
* Age > 18 years
* Adequate performance status of ECOG 0-2
* Life expectancy of at least 3 months
* Written informed consent to participate in the study
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >3,000/uL
  * absolute neutrophil count >1,500/uL
  * platelets >100,000/uL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) < 2.5X normal . Creatinine within normal range and CCT(Cockcroft-Gault) > 50 ml/min

Exclusion Criteria:

* Prior treatment with anti-EGFR or chemotherapy/radiotherapy
* Evidence of CNS metastases
* Poor performance status (ECOG 3-4)
* Evidence of severe or uncontrolled systemic disease (eg. unstable or uncompensated respiratory disorder, cardiac failure, hepatic decompensation, renal failure, nephritic syndrome, uncontrolled metabolic disorders such as diabetes mellitus, uncontrolled hypertension or uncontrolled significant infections)
* Pregnancy or breast-feeding (women of child-bearing potential)
* Prior severe allergic drug reactions
* Prior history of cancer in the last 5 years prior to enrollment, other than curatively treated cancer of the cervix or non-melanoma skin cancer.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04-28 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of locally advanced HNSCC to treatment with Nimotuzumab and concurrent Cisplatin (CDDP) and Radiotherapy (RT). | 16 weeks

SECONDARY OUTCOMES:
To assess the toxicities associated with this regimen | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Teck Lim, MD, Principal Investigator — National Cancer Center Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore